CLINICAL TRIAL: NCT05848401
Title: Biosound Therapy as a Treatment for Long COVID Patients: A Randomized Pilot Trial
Brief Title: Biosound Therapy as a Treatment for Long COVID Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anxiety Relief Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-ANXI-101
Record Dates: First submitted 2023-05-05; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Long COVID
Keywords: long COVID; long haulers; post COVID syndrome; vibroacoustic therapy; biofeedback
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Biofeedback, Psychology

STUDY DESIGN:
Masking Description: Participants were aware they would be placed in the treatment or control group after providing informed consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): The treatment group will be given the following assessments at baseline and four weeks post-randomization: the Patient Health Questionnaire (PHQ-9), Generalized Anxiety Disorder 7-item scale (GAD-7), Cambridge Brain Sciences (CBS) tasks, and the COVID-19 Persistent Symptom Questionnaire. The principal investigator will schedule two Biosound Therapy sessions per week for four weeks for all treatment group participants. The treatment sessions will not occur on consecutive days. All participants in the treatment group will listen to identical playlists. At the beginning of the BTS session, the participant will complete a session of HeartMath biofeedback. Next, the participant will receive approximately 30-40 minutes of music containing binaural beats synchronized with sound massage.The session will finish with gratitude-based video content.
  Interventions: Device: Biosound Therapy System
- Control Group (No Intervention): The control group will be given the following assessments at baseline and four weeks post-randomization: the Patient Health Questionnaire (PHQ-9), Generalized Anxiety Disorder 7-item scale (GAD-7), Cambridge Brain Sciences (CBS) tasks, and the COVID-19 Persistent Symptom Questionnaire. Control group participants were given a complimentary Biosound Therapy session and a ten dollar gift card upon completion of their final assessments.

INTERVENTIONS:
Device: Biosound Therapy System — Biosound Therapy consists of biofeedback, vibroacoustic therapy synchronized with music that plays binaural beats, and video content.
  Other Names: vibroacoustic therapy; biofeedback; binaural beats
  Arms: Treatment Group

SUMMARY:
This study aimed to explore the impact of the Biosound Therapy Systerm on long COVID symptoms while determining feasibility of a future full-scale Randomized Controlled Trial. It was hypothesized that Biosound treatment would significantly improve long COVID.

The goal of this clinical trial is to learn about Biosound Therapy System's impact on long COVID symptoms. The main questions it aims to answer are:

* How does Biosound Therapy impact long COVID symptoms?
* Is the protocol for this trial feasible for a future full-scale Randomized Controlled Trial?

Participants with long COVID symptoms will be assigned to a control group and treatment group. The control group will receive no treatment. The treatment group will have 8 sessions of Biosound Therapy. Researchers will compare the treatment and control group to see if there's a difference in long COVID symptoms.

DETAILED DESCRIPTION:
Investigators will recruit participants through social media and word of mouth. They will also share the study information with practitioners, businesses, organizations, research departments, universities, and the community. Participants will email or call The Anxiety Relief Center to inquire about participating in the study.

Initial screening procedures will take place using the receptionist script to determine eligibility of participants. Eligible participants who agree to participate in the study will then be asked to come into the office for an intake at a time convenient for them. This appointment will include signing the consent form and the completion of initial assessments: Cambridge Brain Sciences tasks, PHQ9, GAD7, and the COVID-19 Persistent Symptom Questionnaire.

After a participant has completed the initial intake appointment, the participant will be randomly assigned to the treatment or control group using Randomizer.org, a computer-generated randomizer. Each participant will be informed if they were assigned to the treatment or control group. An investigator will schedule two Biosound Therapy sessions per week for four weeks with every participant in the treatment group.

The Biosound Therapy System (BTS) is a system that utilizes biofeedback, vibroacoustic technology, and binaural beats. Vibroacoustic Technology uses sinusoidal, low-frequency, rhythmical pulsing sound waves in conjunction with music. The BTS device does not send electricity through the body; rather, the device uses amplifiers embedded into an adjustable bed to send frequencies between 40 and 70 Hz into the body.

At the beginning of the BTS session, the participant will complete the "Biosound Technologies Pretest" questionnaire and then will be instructed to sit on the BTS platform to begin utilizing HeartMath technology that will collect data on heart rate variability (HRV). An investigator will assist the client in attaching a finger sensor around their index finger as they recline onto the platform so that they are facing a monitor positioned in front of the platform. The monitor digitally portrays the participant's HRV and allows the participant to visually see how the rate of their breath is connected to their HRV. The participant spends a few minutes trying to match their breath rate with a moving icon called a breath pacer that is shown on the monitor. The icon moves up and down at the rate of the client's target heart rate. The monitor also displays corresponding coherence levels, which refer to the stability and balance between the brain and nervous system (HeartMath Institute, 2016). The coherence levels are color coordinated with the levels of low, medium, and high. A high coherence level signifies high stability, balance, and regulation, whereas a low coherence level signifies instability, imbalance, and dysregulation. A person with a high coherence level can operate with high efficiency. Once the participant improves their coherence level and HRV (about 5-10 minutes), an investigator will remove the finger sensor and instruct the participant to put on headphones.

Then, an investigator will begin a playlist that includes music with binaural beats that is synchronized with sound massage. Once the playlist has begun, an investigator will turn off the lights and exit the room until the playlist is finished. The session ends with video content. Each participant will be given an identical playlist for each session. At the end of the session, the participant will complete the "Biosound Technologies Posttest" questionnaire to assess the perceived effects of the session.

All collected data will be deidentified and stored in a HIPAA compliant electronic medical record system called Therapy Appointment. After a participant in the treatment group has completed their treatment sessions, they will complete the same assessments given at intake. After the assessments are completed, an investigator will ask 2 open-ended questions and then will record a summary of their answers.

While Biosound Therapy rarely causes side effects, some people may experience dizziness or discomfort. While adverse reactions are rarely reported, a decreased sense of anxiety can feel unfamiliar to people who are used to a state of physiological increased awareness. As stated above, the BTS is a wellness device that was designed to provide relief and side effects are rarely reported. All participants will be told that they can stop treatment at any time during the session by leaving the treatment room. An investigator will be in close proximity to the treatment room at all times to provide any needed assistance during participants' sessions. Snacks, water, guidance and emotional support will be available to participants should they experience any side effects. Additionally, HRV allows subjects an opportunity to see a balanced and healthy state and can help center a client who may be feeling dizzy after sound massage. The investigators will record any adverse side effects reported by the participants.

The process measures of recruitment and retention rates, open-ended interview responses, and participant characteristics will be summarized using descriptive statistics. Due to the small sample size, the Wilcoxon signed-rank test will be used to determine changes in the variables for the intervention and control group.

ELIGIBILITY:
Inclusion Criteria:

* experiencing at least three symptoms that began or were intensified due to COVID
* able to provide documentation of a COVID-19 test older than 30 days.
* 20-65 years old.

Exclusion Criteria:

* abusing alcohol or drugs
* having a pacemaker or any other implanted devices
* pregnancy
* history of the following conditions: blood clots, schizophrenia, seizures, recent head injury, and any acute physical injury

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
The Patient Health Questionnaire (PHQ-9) | 4 weeks
  9-item questionnaire assessing for Major Depressive Disorder
Generalized Anxiety Disorder 7-item scale (GAD-7) | 4 weeks
  7-item questionnaire assessing for generalized anxiety disorder
Cambridge Brain Sciences (CBS) tasks | 4 weeks
  The CBS tasks measure reasoning, short-term memory, and verbal ability through 12 online tasks simulating puzzles or video games.
COVID-19 Persistent Symptom Questionnaire. | 4 weeks
  The authors developed The COVID-19 Persistent Symptom Questionnaire to measure common persistent COVID-19 symptoms at their worst over the last week on a scale of 0-3.

SECONDARY OUTCOMES:
Recruitment Rate | Through study completion, an average of 1 year
  Recruiting individuals with long COVID symptoms into a trial of the Biosound Therapy System
Retention Rate | 4 weeks
  Retaining participants for a 4 week trial for the proposed battery of assessments. Retention rate (%) of participants enrolled into the trial who completed the 4 week protocol.
Open-ended questions to participants about their experience | 4 weeks
  Participants will be asked, "1. Can you describe your experience receiving BTS in this study? 2. How did you perceive this treatment helping or not helping your symptoms?"

CONTACTS AND LOCATIONS:
Overall Officials: Colleenia R Korapatti, MA, Principal Investigator
Locations (1):
- The Anxiety Relief Center, Fishers, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Any researchers who are interested in replicating the study or using the de-identified IPD can contact the principal investigator for a copy of the data set.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available indefinitely after the completion of the study.
Access Criteria: The principal investigator Colleenia Korapatti will review requests upon contact. Requested information will be shared electronically.